CLINICAL TRIAL: NCT02494882
Title: Phase I Trial Adding Ruxolitinib to a Combination of Dasatinib Plus Dexamethasone in Remission Induction Therapy in Newly Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia Patients Aged 40 Years or Older.
Brief Title: Adding Ruxolitinib to a Combination of Dasatinib Plus Dexamethasone in Remission Induction Therapy in Newly Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia Patients Aged 40 Years or Older
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Incyte Corporation (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-272
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Ruxolitinib; Dasatinib; Dexamethasone; 14-272
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ruxolitinib; Dasatinib; Dexamethasone

ARMS (1):
- Adding Ruxolitinib to Combination of Dasatinib + Dexamethasone (Experimental): Steroid Pre-Phase (Days -6 to 0) Prednisone 10 mg/m2/day uptitrated to 60/mg/m2/day oral over seven days (capped at 120 mg/day).
  Remission Induction (Days 1 to 84) Dasatinib 140 mg oral once daily. Days 1-84. Dexamethasone 10 mg/m2/day oral (capped at 20 mg/day). Days 1-24. Dexamethasone oral taper 10 mg/m2/day (capped at 20 mg/day) to off. Taper days 25-32. Off day 33.
  Ruxolitinib phase I cohort dose oral. Days 1-84. Delivered BID. Delivered per the phase I dose cohort. Methotrexate (MTX) 12 mg Intrathecal (IT) for 4 doses on days 22, 43, 64, 85; +/- 3 days.
  Post-Remission Induction Therapy (Starting Day 85) Allogeneic HSCT, at the discretion of the treating physician, at any point post-remission induction.
  Or, post-remission induction (consolidation) therapy to be determined per the treating physician
  Interventions: Drug: Ruxolitinib; Drug: Dasatinib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ruxolitinib
Drug: Dasatinib
Drug: Dexamethasone

SUMMARY:
The purpose of this study is to test the safety of a new combination of three oral drugs in Ph+ ALL. These drugs are dexamethasone, dasatinib, and ruxolitinib. All three drugs have been studied before in humans.

This is a phase I study in which ruxolitinib dose will start low for the first patient together with dexamethasone plus dasatinib. If this dose does not cause a bad side effect, the ruxolitinib dose will slowly be made higher as new patients take part in the study. This will help the investigators find the right dose of ruxolitinib to give together with dexamethasone and dasatinib that will be used in future studies

ELIGIBILITY:
Inclusion Criteria:

* Patient able to give informed consent.
* Patients >/= 18 years with the following disease will be eligible

  * Newly diagnosed Ph+ ALL, previously untreated, except for the below allowances
  * Previously received HpyerCVAD cycle 1A+/- cycle 1B
  * Previously received Induction Phase 1 +/- Induction Phase II of BFM-modeled (Pediatric of Pediatric-Inspired) ALL regimen
  * Previously received other representative (modified from HyperCVAD, BFM, or AML-like) ALL induction course, including ABL TKI plus corticosteroid.
  * If the patient has received any of the above prior therapy, they may be enrolled, regardless of remission status.
  * Relapsed PH+ ALL, with no prior exposure to dasatinib and without known ABL kinase mutations predited to be resistant to dasatibin (e.g. L248R, L248V, Q252H, E255K, V299L, T315A, T315I, F317C, F317L, F317S, F317V)
  * Relapsed or refractory Ph-like ALL without prior exposure to dasatibin and with mutations or rearrangements of genes conferring sensitivity to dasatibin (ABL, CSF1R, PDGFRB) or ruxolitinib (CRLF2, JAK3, EPOR, TSLP)
  * Newly diagnosed or relapsed CML in lymphoid blast crisis
* Confirmation of Philadelphia chromosome positivity by cytogenetics (karyotype/FISH) and/or molecular tests (BCR-ABL1 transcripts)
* Acceptable end-organ function, except for documented exclusions for organ function compromise due to ALL itself
* ECOG performance status ≤ 2
* Men and women of childbearing potential must be willing to practice an effective method of birth control during treatment and for at least 4 months following treatment on study

Exclusion Criteria:

* Ph-negative ALL
* Patients with dominant leukemic clone bearing documented bcr-abl mutations enabling bcr-abl TKI resistance at diagnosis
* Mature B-cell (Burkitt's) ALL
* Serum creatinine > 1.5x ULN and calculated creatinine clearance, based on a 24-hour urine collection, < 30 mL/min--unless related to ALL/tumor lysis syndrome and able to be corrected
* Direct Bilirubin > 2x ULN; AST/ALT > 10x ULN, unless related to ALL liver infiltration.
* Pregnant women or women who are breast-feeding
* Patients with HIV, Hepatitis B, or Hepatitis C
* Pre-treatment QTcF > 480 msecs
* A "washout" period of at least 14 days from last previous cytotoxic chemotherapy will be required prior to starting treatment on this protocol. No "washout" period will be required for previous bcr-abl TKI therapy given with the aforementioned previous chemotherapy cycles. Hydroxyurea and corticosteroids may be given as bridge therapy up until 24 hours prior to initiating protocol treatment.
* Active malignancy requiring treatment other than ALL within two years prior to start of treatment, with the exception of basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, localized prostate cancer, or DCIS or LCIS of the breast
* Active, uncontrolled infection, any other concurrent disease, or medical condition that is deemed to interfere with the conduct of the study as judged by the investigator
* Unable to tolerate anti-viral and anti- Pneumocystis jirovecii prophylaxis while on pre-phase and remission induction therapy
* Unable to tolerate gastrointestinal prophylaxis therapy with sucralfate while on pre-phase and remission induction therapy. Or severe pre-existing GI disorder that requires PPI or H2 receptor antagonist therapy be uninterrupted

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical response | 2 years
  is to be evaluated by using a combination of criteria. Molecular remissions will be defined by standard criteria for BCR-ABL1 and IGH qRT-PCR. Flow cytometric assessment of MRD will be defined by standard flow cytometry criteria

SECONDARY OUTCOMES:
Complete Molecular Remission (CMR) rate | 2 years
  Molecular remission status will be defined by undetectable BCR-ABL1 transcripts and/or IGH clonal gene rearrangement in bone marrow aspirate (BMA) examination as determined by qRT-PCR in CLIA laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/